CLINICAL TRIAL: NCT06643039
Title: Hospital-acquired Respiratory Viral Infection: A Prospective Multicenter Study in France
Brief Title: Nosocomial Respiratory Virus Infection
Acronym: NOSOVIRUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL23_1091; 2024-A01267-40 (Other: ID-RCB)
Record Dates: First submitted 2024-10-14; First posted 2024-10-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Nosocomial Infections
Keywords: Hospital-acquired infection; COVID-19; Influenza; SRV; France
MeSH Terms: conditions — Cross Infection; COVID-19; Influenza, Human | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients hospitalized in participating services for more than 24h (Other): Patients hospitalized for more than 24 hours in the participating services (geriatric, internal medicine, transplantation) and who presents an influenza like illness (ILI) on admission or during hospital stay are eligible to participate. Following the signature of the consent, nasopharyngeal sample will be collected. Socio-demographic (questionnaire) and clinical information will be obtained using the study e-CRF.
  Interventions: Biological: Nasopharyngeal swab; Other: Questionnaire
- Volunteered health care professionals (Other): Volunteered health care professionals in the participating services (geriatric, internal medicine, transplantation) and who presents an influenza like illness (ILI) are eligible to participate. Following the signature of the consent, nasopharyngeal sample will be collected. Socio-demographic (questionnaire) and clinical information will be obtained using the study e-CRF
  Interventions: Biological: Nasopharyngeal swab; Other: Questionnaire

INTERVENTIONS:
Biological: Nasopharyngeal swab — Nasopharyngeal swab collection will be carried out in patients and health care professionals presenting an ILI during the study period. This will be done by trained clinical research associates after the signature of the consent. Only one nasopharyngeal sample is expected to be collected from each participant.
Other: Questionnaire — questionnaire including demographic data, data on medical history and vaccination, and clinical and biological data on the viral episode.

SUMMARY:
Hospital-acquired Viral Respiratory Infections (HAVRI) are associated with substantial burden on health care systems. The prevention and control of these viral infections rely on multiple measures such as hand hygiene or wearing mask. However, vaccination remains the major preventive measure.

To date, data at French national level are insufficient to describe the epidemiology of these infections, including their burden, and the potential protection of patients if vaccination coverage of health care professionals/patients is satisfactory. In addition, better understanding of the clinical characteristics of HAVRI will make it possible to identify potential sources of transmission as soon as possible and to implement appropriate hygiene measures.

We will set up a hospital-based prospective multicenter study in Bordeaux, Paris-Bichat, Dijon and Lyon, involving four inclusion services (geriatrics, internal medicine and transplantation) per hospital.

The main objective of this study is to calculate the incidence rate of hospital-acquired infections for three respiratory viruses; influenza, SARS-CoV-2 and syncytial respiratory virus (SRV), referred to as HARVI, in participating services.

Volunteered health care professionals or hospitalized patients presenting with influenza-like illness (ILI) at admission or during their stay in the participating centers will be eligible to be enrolled during the two inclusion periods: (mid-October 2024 to mid-April 2025 and mid-October 2025 to mid-April 2026).

For each patient/health care professional, a nasopharyngeal swab will be collected. A questionnaire including demographic data, medical history, vaccination, and clinical and biological data of the viral episode will also be completed by the study team. Patients tested positive for one of the viruses studied will be considered "cases" and patients tested negative as "controls".

The collected data will be pseudonymized before statistical analyses. Statistical analyses will consist of calculating incidence rates, attack rates overall and by causative virus and analysis of factors associated with the occurrence of HARVI.

The prospective design of the study will optimize the quality of the collected data (ex. consolidate the documentation of both the clinical picture and vaccination in patients and health care professionals by reducing memory bias) and allow to calculate the incidence rates, the crude and adjusted relative risks of HARVI according to the studied factors, and to describe multiple outcomes (hospitalization in intensive care units, death, etc.) based on the causative virus.

The results of this research project will allow to:

* obtain epidemiological indicators associated with HARVI;
* estimate the impact of HARVI on the prognosis of patients in hospital;
* assess the impact of HARVI on the total length of hospital stay;
* identify risk factors associated with HARVI;
* use the results as an argument for vaccination in order to increase vaccination coverage of healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Adults> 18 years old
* Hospitalized patient or health care professionals presenting an ILI on admission or during the stay, meeting the following definition: fever greater than 37.8° C in the absence of taking antipyretics and/or cough or pharyngeal pain.
* Signed consent form

Exclusion Criteria:

* Pregnant, parturient or breastfeeding women
* individuals deprived of their liberty by a judicial or administrative decision
* Individuals subject to psychiatric care
* Individuals admitted to a health or social establishment for purposes other than research
* Individuals under a legal protection measure (guardianship, curatorship)
* Individuals not affiliated to a social security insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of hospital-acquired respiratory viral infections | At inclusion
  The primary endpoint will be evaluated by calculating the incidence of hospital-acquired respiratory viral infections overall and by type of virus (influenza, COVID-19, RSV) during the surveillance period.
  incidence rate will be estimated by the ration of number of incident cases over the study period to the cumulative observation time (in person-weeks) of hospitalized patients.
  Incidence density will be estimated by the ratio of number of incident cases during successive weekly observation periods to the cumulative observation times calculated over the same periods.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Pellegrin Hospital, Bordeaux
  - CHU Dijon, Dijon
  - Edouard Herriot Hospital, Lyon
  - Bichat Hospital, Paris